CLINICAL TRIAL: NCT04960358
Title: The Application Of Surface Electromyography (SEMG) In Stratifying Chronic Low Back Pain
Brief Title: Surface Electromyography in Stratifying Chronic Low Back Pain.
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Anwar Suhaimi, Dr, University of Malaya
Other Study IDs: 201948-7312
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic LBP: Will be applied Surface Electromyography
  Interventions: Procedure: Surface Electromyography

INTERVENTIONS:
Procedure: Surface Electromyography — will be applied Surface Electromyography to assess Flexion Relaxation Response

SUMMARY:
Surface Electromyography can be utilised to detect normal muscle electrical activity during maximum forward flexion termed Flexion Relaxation Response (FRR)

DETAILED DESCRIPTION:
In this study, our primary objective is to assess FRR and disability (ODI) correlation protocol as an objective tool in stratifying Chronic LBP. We also would like to evaluate the relationship between FRR with pain intensity and lumbar range of motion as our secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 20 - 70 years old
* Mechanical LBP > 6 weeks (not acute LBP)
* Not received any specific exercise spinal manipulation or surgery to improve LBP within the last 3 months.

Exclusion Criteria:

* Pregnancy
* Radicular LBP patients or specific-spinal pathology / "red-flags".
* Surgical intervention for the current LBP complaint (includes traumatic causes of LBP with surgical intervention)
* Cognitive or communication difficulty preventing active participation in exercises or communicating pain scores

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain who were being referred to the rehabilitation outpatient in University Malaya Medical Centre between November 2019 until July 2020.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 1 YEAR
  Questionnaire of the functional assessment for the low back pain patient
Flexion Relaxation Response (FRR) ratio | 1 YEAR
  The FRR ratio was calculated from the best SEMG values obtained during Forward Lumbar Flexion & Extension

SECONDARY OUTCOMES:
Visual Analog Scale | 1 YEAR
  Representing range of pain intensity from no pain on the far left to most intense pain on the far right.
Gross Range of Motion | 1 YEAR
  Degree of trunk motion at maximum voluntary flexion, measured by inclinometer at the level of T12

CONTACTS AND LOCATIONS:
Overall Officials: ANWAR SUHAIMI, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided